CLINICAL TRIAL: NCT06474442
Title: A Multicenter, Single-blind, Single-dose, Randomized, Phase Ⅱa Trial to Evaluate the Safety, Tolerability and Efficacy of Intrastromal BD111 Gene Editing Therapy in Adults With HSV-1 Stromal Keratitis
Brief Title: A Phase Ⅱa Study of the Safety, Tolerability and Efficacy of BD111 in Herpes Simplex Virus Type I Stromal Keratitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BD-HSK-111002-Ⅱa
Record Dates: First submitted 2024-06-13; First posted 2024-06-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Herpes Simplex Virus Type I Stromal Keratitis
Keywords: Herpes Simplex Virus Type I; Stromal Keratitis
MeSH Terms: interventions — Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): BD111 combining triple-drugs therapy Group.
  Interventions: Genetic: BD111 Injection (investigational new drug); Combination Product: Triple-drugs therapy of HSV-1 stromal keratitis
- Group 2 (Active Comparator): BD111 sham injection combining triple-drugs therapy group.
  Interventions: Combination Product: Triple-drugs therapy of HSV-1 stromal keratitis

INTERVENTIONS:
Genetic: BD111 Injection (investigational new drug) — BD111: intrastromally injection, single-dosing 10E6 TU/eye, specified injection volume is 0.15mL.
  Other Names: BD111 Lentivirus-like particles, also called HSV-1-erasing lentiviral particles (HELP)
  Arms: Group 1
Combination Product: Triple-drugs therapy of HSV-1 stromal keratitis — Triple-drugs therapy: "Ganciclovir Eye gel+Valacilovir Tablets+Prednisolone Acetate Eye Drops" for 3 weeks.
  Other Names: Ganciclovir Eye gel+Valacilovir Tablets+Prednisolone Acetate Eye Drops

SUMMARY:
This study aims to compare the clinical efficacy and safety of BD111 injection in combination with standard therapy vs. standard therapy in herpes simplex virus type I stromal keratitis (HSK), providing preliminary confirmation of the clinical effectiveness of BD111 in combination with standard therapy.

DETAILED DESCRIPTION:
This is a phase Ⅱa, single-blind, single-dose, randomized, positively controlled clinical trial of BD111 in patients with herpes simplex virus type I stromal keratitis (HSK) aged 18 to 70 years. Forty eligible participants will be recruited in the trial. BD111 is investigational new biologics (Injection)--a type of lentiviral-like particle that can simultaneously deliver SpCas9 and gRNA targeting the HSV-1 virus gene, also known as HSV-1-erasing lentiviral particles (HELP). The total follow-up duration was 12 months, the safe endpoints and efficacy endpoints will be used to assess the efficacy, safety and tolerability profiles in patients with HSK.

ELIGIBILITY:
Inclusion Criteria: Participants must meet all of the following inclusion criteria to be enrolled in this study.

1. Aged 18 to 70 years old;
2. Clinically diagnosed with herpes simplex virus stromal keratitis;
3. Tear swab HSV-1 nucleic acid test (qPCR method) positive;
4. No use of systemic antiviral drugs or corticosteroids within 48 hours before enrollment;
5. No systemic immune eye diseases;
6. Good eyelid structure and blinking function;
7. Eye structure and function assessment showing potential for visual recovery;
8. No retinal detachment, with generally normal visual function;
9. No history of corneal trauma;
10. Visual acuity in the fellow eye is better than 20/200;
11. Fertile males or females must use highly effective contraceptive methods (such as oral contraceptives, intrauterine devices, abstinence, or barrier contraception combined with spermicides) during the trial and continue contraception for 12 months after administration;
12. Participants voluntarily join the study, sign an informed consent form, have good compliance, and cooperate with follow-up visits.

Exclusion Criteria: Patients with any of the following conditions cannot be enrolled in this study

1. Active ocular infection caused by other pathogens in the target eye or the fellow eye within 30 days before enrollment, including but not limited to blepharitis, infectious conjunctivitis, keratitis, scleritis, and endophthalmitis;
2. Patients with bilateral viral keratitis
3. Previous corneal transplant surgery in the study eye;
4. A history of adverse reactions or allergies to corticosteroids and sodium fluorescein, allergies to therapeutic or diagnostic protein products, allergies to ≥ two drugs or non-drug factors, or having an ongoing allergic disease;
5. Absence of tear film and blinking function;
6. Severe dry eye disease;
7. Malignant ocular surface tumor;
8. Glaucoma;
9. Patients with systemic autoimmune diseases;
10. Signs of systemic infection before enrollment, including fever and receiving antibiotic treatment (abnormal elevating values in white blood cells, lymphocytes, and neutrophils in routine blood tests);
11. Abnormal major organ function or other uncontrolled clinical problems, mainly including but not limited to the following:

    * Severe kidney disease history, serum creatinine ≥ 133μmol/L;
    * Liver dysfunction, transaminase level ≥ 80 IU/L;
    * Uncontrolled hypertension, systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg;
    * Uncontrolled diabetes, fasting blood glucose greater than or equal to 8.0 μmol/L;
    * Cardiovascular disease history, with arrhythmia, myocardial ischemia, and myocardial infarction (diagnosed by electrocardiogram examination);
    * Platelet level ≤ 100×10^9/μL or ≥ 450×10^9/μL due to any cause, hemoglobin level lower than 10.0g/dL (male) or 9.0g/dL (female).
12. HIV infection;
13. Pregnant and lactating women (pregnancy in this trial is defined as a positive urine pregnancy test);
14. Participation in other drug or medical device clinical trials;
15. Alcohol or drug abuse;
16. Lack of compliance with the trial or the ability to sign an informed consent form;
17. Other situations deemed unsuitable for participation in the trial by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate of HSK at Day 70 and Day112 post-administration | 12 months
  Definition of HSK clinical cure: disappearance of the subject's clinical symptoms, disappearance of active inflammatory lesions on ophthalmologic examinations, and successful clearance of the HSV-1 viral genome.

SECONDARY OUTCOMES:
The percentage of participants with successful clearance of HSV-1 viral genome in tears at Day 14, Day 28, Day 70, Day 112, Day 180, and Day 365 post-administration | 12 months
  The definition of successful HSV-1 clearance: negative results in tear swab HSV-1 nucleic acid tests on two consecutive samplings (interval ≥14 days).
  The definition of a negative result in tear swab HSV-1 nucleic acid test: single qPCR Ct value = 40 or "undetected", or Ct value of the first qPCR test "36 < Ct value < 40", and the Ct value of repetitive qPCR test is 40 or "undetected".
The percentage of participants with failed clearance of HSV-1 viral genome in tears at Day 14, Day 28, Day 70, Day 112, Day 180, and Day 365 post-administration | 12 months
  The failure of HSV-1 viral genome clearance is determinated by HSV-1 positive results of qPCR test. HSV-1 positive definition of qPCR test: qPCR Ct value ≤ 36, or qPCR Ct value is "36 < Ct value < 40" and the Ct value of repetitive qPCR test is ≤ 36, or results of both qPCR tests are "36 < Ct value < 40".
The percentage of participants with HSK recurrence at Day 180, and Day 365 post-administration | 12 months
  Definition of HSK recurrence: HSV-1 nucleic acid qPCR test is positive, and clinical symptoms presents again, and ophthalmic examinations find active inflammatory lesions on interventional eye.
Score change of corneal inflammation scale post-administration | 12 months
  From baseline to Day 70, Day 112, Day 180, and Day 365 post-administration.
The improvement in best corrected visual acuity (BCVA) | 12 months
  From baseline to Day 70, Day 112, Day 180, and Day 365 post-administration.
The improvement in corrected distance visual acuity (CDVA) post-administration | 12 months
  From baseline to Day 70, D11ay 2, Day 180, and Day 365 post-administration.
Anti-p24 antibody in blood | 12 months
  At Day 14, Day 28, Day 112, Day 180, and Day 365 post-administration.
Anti-Cas9 antibody in blood | 12 months
  At Day 14, Day 28, Day 112, Day 180, and Day 365 post-administration.
Anti-BD111 antibody in blood | 12 months
  At Day 14, Day 28, Day 112, Day 180, and Day 365 post-administration.
Vector RNA copy number in tear fluid | 12 months
  Vector persistence times: Tear fluid vector RNA copy number at Day 112, Day 180, and Day 365 post-administration.
Circular DNA copy number in blood | 12 months
  Vector persistence times: circular DNA copy number in blood at Day 112, Day 180, and Day 365 post-administration.
Off-target Detection | 6 months
  BD111 off-target detection (DNA deep sequencing) in eye swabs at Day 14 and Day 180 post-administration
The characteristics of adverse events (AEs) and serious adverse events (SAEs) | 12 months
  AEs and SAEs are recorded and evaluated (type, incidance, severity etc.), including ocular and systemic AEs/SAEs post-administration.

CONTACTS AND LOCATIONS:
Overall Officials: Fujun Li, M.D., Study Director — Shanghai BDgene Co., Ltd.
Locations (1):
- Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China